CLINICAL TRIAL: NCT05905120
Title: A Single-Arm, Non-Randomized, Open-Label, Exploratory Mechanistic Validation (PoM) Clinical Trial of Toludivenlafaxine Hydrochloride Extended-Release Tablets Assessing Dopamine Transporter Occupancy in the Healthy Adult Brain Using 11C-CFT Positron Emission Tomography (PET)
Brief Title: Assessing Dopamine Transporter Occupancy in the Healthy Adult Brain With Toludivenlafaxine Hydrochloride Extended-Release Tablets Using 11C-CFT Positron Emission Tomography (PET)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Yantai University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMHC-224
Record Dates: First submitted 2023-06-01; First posted 2023-06-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toludivenlafaxine hydrochloride sustained-release tablets (Experimental): 80 mg/tablet, 2 tablets each time, once a day, for 4 days
  Interventions: Drug: Toludivenlafaxine hydrochloride sustained-release tablets

INTERVENTIONS:
Drug: Toludivenlafaxine hydrochloride sustained-release tablets — 80 mg/tablet, 2 tablets each time, once a day, for 4 days, orally at 30 min after the start of meals, 200 mL water to take

SUMMARY:
This study was a single-arm, non-randomized, open-label clinical study to assess dopamine transporter occupancy in the brain of healthy adults using 11C-CFT positron emission tomography (PET)

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily participate in and sign the informed consent form after understanding the purpose, content, process and possible risks of the trial;
2. Male, aged 18 to 45 years at the time of signing the informed consent form;
3. Body weight ≥ 50.0 kg and body mass index (BMI) 18.5 ~ 28.0 kg/m2 (including the boundary value) at screening;
4. Able to maintain good communication with the investigator and comply with the lifestyle restrictions specified in the protocol and various requirements of the clinical trial (scheduled visits, laboratory tests and other trial procedures);
5. Male subjects and their partners must use effective non-pharmacological contraception (e.g., abstinence and condom with intravaginal spermicide) throughout the study and for 6 months after the end of the study, and must not donate sperm.

Exclusion Criteria:

1. Known to have a history of allergy to any component of the investigational product or similar drugs, or allergic constitution (previous allergy to two or more foods or drugs);
2. The subject has a current or past medical history judged by the investigator that may affect the clinical trial or dysfunction, including but not limited to a past or present respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, motor system, blood system, psychiatry, dermatology and any other clinically significant disease or chronic disease; or any other disease that may interfere with the test results;
3. Any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects participating in the trial; such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, gastrointestinal bleeding, etc.;
4. Abnormal vital signs, laboratory tests, 12 electrocardiogram (ECG), MRI (magnetic resonance imaging) examination indicators, judged by the investigator as abnormal and clinically significant;
5. Use of the following medications or treatments prior to dosing:

   Use of any prescription medication within 28 days prior to dosing; Use of any over-the-counter medications, including health products, within 7 days prior to dosing; Receipt of any contrast agent or radiopharmaceutical within 48 hours prior to, or application of contrast agent within 24 hours after, administration of the trial drug;
6. Contraindications to PET or MRI (magnetic resonance imaging) (including claustrophobia, alcohol allergy, cardiac pacemaker and nerve stimulator in the body, metal foreign body in the body or tracer component allergy, etc.);
7. Any positive result of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab) and tolulized red unheated serum test (Trust);
8. Smoking habit (an average daily smoking of ≥ 5 cigarettes per day within 3 months before administration), drinking habit (an average weekly drinking of more than 14 standard units within 3 months before administration, 1 unit = 360 mL of beer or 45 mL of 40% spirits or 150 mL of wine), history of drug abuse or positive results of urine drug screening;
9. Those who have special requirements for food and cannot abide by the unified diet or have dysphagia;
10. Consumption of xanthine-rich foods or beverages (e.g., tea, coffee, cola, or chocolate) or foods or beverages containing grapefruit and/or pomelo within 3 days before dosing;
11. Significant occupational exposure to ionizing radiation (e.g., more than 50 millivolts per year) or exposure to radioactive substances or ionizing radiation for therapeutic or research purposes within the past 10 years;
12. Blood donation or blood loss ≥ 400 mL within 3 months before administration, or blood donation or blood loss ≥ 200 mL within one month;
13. Those who have participated in other clinical trials within 3 months before administration (including drug and medical device clinical trials, the time is based on the last visit, except for those who have failed screening in other clinical trials and have not received any treatment);
14. Have a history of suitable to participate in the study as judged by the investigator;
15. Personnel directly related to this clinical trial;
16. Patients with poor compliance or other problems who are not suitable for participating in this trial in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Dopamine Transporters Occupancy in the Basal Ganglia（Positron emission tomography with 11C-CFT was determine by SUVr of the Basal Ganglia DAT） in Human Brain by Toludivenlafaxine Hydrochloride Extended-Release Tablets | from baseline to day 4

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng SHEN, MD, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No